CLINICAL TRIAL: NCT00968604
Title: A Phase I Open-Label Dose Escalation Study to Assess the Safety and Tolerability of the BikDD Nanoparticle in Patients With Advanced Pancreatic Cancer
Brief Title: C-VISA BikDD: Liposome in Advanced Pancreatic Cancer
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Stability of the DNA when admixed with the liposome failed
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2007-0762; 1 R21 CA135 60401A1 (Other Grant/Funding Number: NCI); NCI-2011-00466 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2009-08-28; First posted 2009-08-31 (Estimated); Last update posted 2019-04-11 (Actual); Status verified 2019-04

CONDITIONS: Pancreatic Cancer
Keywords: Pancreatic Cancer; Pancreas; Liver; Liver Tumor Biopsy; BikDD Nanoparticle; C-VISA BikDD
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- BikDD Nanoparticle (Experimental): BikDD Nanoparticle starting dose 0.04 mg/kg once weekly by vein over 10 minutes.
  Interventions: Genetic: BikDD Nanoparticle

INTERVENTIONS:
Genetic: BikDD Nanoparticle — Starting dose 0.04 mg/kg once weekly by vein over 10 minutes.
  Other Names: Bik gene product; Cholesterol liposome-based nanoparticle

SUMMARY:
The goal of this clinical research study is to find the highest tolerable dose of BikDD nanoparticle that can be given to patients with advanced cancer of the pancreas. The safety of this drug will also be studied.

DETAILED DESCRIPTION:
The Study Drug:

BikDD is a modified gene product that is designed to make cancer cells destroy themselves. Delivering BikDD in a fat molecule (a BikDD nanoparticle) may improve the delivery of the gene product into the cells. This may help to stop or slow the growth of pancreatic cancer. This is the first study using BikDD nanoparticle in humans.

Study Drug Dose Level:

If you are found to be eligible to take part in this study, you will be assigned to a dose level of BikDD nanoparticle based on when you joined this study. Different dose levels of BikDD nanoparticle will be tested. Three (3) participants will be enrolled at each dose level. The first group of participants will receive a low dose level. Each new group will receive a higher dose level, if no intolerable side effects were seen. If intolerable side effects were seen, then the next group of participants will receive a lower dose. This will continue until the highest tolerable dose of BikDD nanoparticle is found.

The dose of study drug that you receive will never be increased. However, if you have side effects, your dose of study drug may be lowered. Your doctor will discuss with you which dose you will receive.

Study Drug Administration:

There will be 28 days in each cycle. The study visit schedule is described below. In certain circumstances, with the permission of your doctor, the study visits may occur up to 2 or 3 days earlier or later than described below.

On Days 1, 8, 15, 22 of each cycle, you will receive BikDD nanoparticle through a needle in your vein over about 10 minutes.

Study Visits:

Liver Tumor Biopsy:

Before you receive the study drug, you will have a biopsy of the liver tumor. Researchers will compare this biopsy with a later biopsy to learn if the BikDD nanoparticle will be able to reach the tumor and what effect it is having on the cancer.

You will be awake during the biopsy. A radiologist will find the tumor with the help of a scan such as an ultrasound or CT scan. You will receive a local anesthetic. A needle will be inserted through the skin into the tumor, and tissue sample(s) will be taken. You will receive fluids and drugs for relaxation and/or pain as needed through a needle in your arm or hand.

On Days 1, 8, 15, 22 of Cycle 1, the following tests and procedures will be performed:

* You will have a physical exam, including measurement of your weight.
* Your vital signs will be measured 5 times.
* Your performance status will be recorded.
* You will be asked about any drugs and/or supplements you are taking or have taken since your last visit.
* You will be asked about any side effects you may be experiencing.
* Blood (about 2-3 tablespoons) will be drawn for routine tests.
* On Day 1 only, blood (about 2 teaspoons each time) will be drawn 9 times for pharmacokinetic (PK) testing. PK testing measures the amount of study drug in the body at different time points.

On Day 2 of Cycle 1, blood (about 2 teaspoons) will be drawn 1 time for PK testing.

On Days 4, 11, 18, and 25 of Cycle 1, the following tests and procedures will be performed:

* Blood (about 2-3 tablespoons) will be drawn for routine tests.
* You will be asked about any side effects you may be having.

On Day 24 of Cycle 1, you will have a biopsy of the liver tumor to learn if BikDD nanoparticle is reaching the tumor and its effect on cancer. If for any reason the biopsy can't be performed then, you may be asked to have the biopsy 6-8 days later.

On Day 1 of Cycle 2, the following tests and procedures will be performed:

Your medical history will be recorded, including any drugs and/or supplements you are taking or have taken since your last visit.

* You will have a physical exam, including measurement of your weight.
* Your vital signs will be measured 5 times.
* Your performance status will be recorded.
* You will be asked about any side effects you may be experiencing.
* Blood (about 2-3 tablespoons) and urine will be collected for routine tests.
* You will have an ECG.

On Days 8, 15, and 22 of Cycle 2, the following tests and procedures will be performed:

* Blood (about 1 tablespoon) will be drawn for routine tests.
* Your vital signs will be measured 5 times.
* You will be asked about any side effects you may be experiencing.

At the end of Cycle 2 and every other cycle (Cycle 4, 6, 8, and so on), you will have a CT scan or MRI of the chest, abdomen, and pelvis to check the status of the disease. Blood (about 1 teaspoon) will be drawn to measure your CA 19-9 level. Because it may take some time for the effects BikDD may have on the tumor to be known, the study doctor may decide to continue the BikDD even if the scan/MRI shows the tumor is worse. In this case, you will have another CT scan or MRI of the chest, abdomen, and pelvis 4 to 6 weeks later. If the cancer is worse, you will stop BikDD.

On Day 1 of Cycles 3 and beyond, the following tests and procedures will be performed:

* Your medical history will be recorded, including any drugs and/or supplements you are taking or have taken since your last visit.
* You will have a physical exam, including measurement of your weight.
* Your vital signs will be measured 5 times.
* Your performance status will be recorded.
* You will be asked about any side effects you may be experiencing.
* You will have an ECG.
* Blood (about 2-3 tablespoons) and urine will be collected for routine tests.

On Days 8, 15, and 22 of Cycles 3 and beyond, the following tests and procedures will be performed:

* Your vital signs will be measured 5 times.
* You will be asked about any side effects you may be experiencing.
* Blood (about 2-3 tablespoons) will be drawn for routine tests.

Length of Study:

You may continue to receive the study drug as long as your doctor thinks it is in your best interest. If all of the cancer disappears, you will receive 2 extra cycles of study drug and then stop study drug. You will be taken off study if the disease gets worse, your doctor decides that it is in your best interest to stop the drug, or if you experience intolerable side effects.

End-of-Study Visit:

Once you stop the study drug for any reason, you will have an end-of-study visit. At this visit, the following tests and procedures will be performed.

* Your medical history will be recorded, including any drugs and/or supplements you are taking or have taken since your last visit.
* You will have a physical exam, including measurement of your weight and vital signs
* Your performance status will be recorded.
* You will be asked about any side effects you may be experiencing.
* You will have an ECG.
* Blood (about 2-3 tablespoons) and urine will be collected for routine tests and to measure your CA 19-9 level.
* If you have not had one within the last 4 weeks, you will have a CT scan or MRI of the chest, abdomen, and pelvis to check the status of the disease

Once a week for at least 30 days after your last dose of study drug, you will be asked if you are experiencing any side effects. If you do not have a clinic visit already scheduled, you will be called. If you are called, it will take about 5-10 minutes.

If you experience any side effects, you may continue follow-up visits until the medical problem has gone away or stabilized.

Follow-Up:

Every 2 months from then on, the study staff will continue to see how you are doing, either at a routine clinic visit or by phone. If you are called, it will last about 5-10 minutes. If you move, you will also be asked to provide your new address and telephone number to your doctor.

This is an investigational study. BikDD nanoparticle is not FDA approved or commercially available. At this time, BikDD nanoparticle is only being used in research.

Up to 30 patients will take part in this study. All will be enrolled at M D Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have histologically or cytologically confirmed advanced pancreatic adenocarcinoma that is unresectable or metastatic.
2. Patient must have received prior gemcitabine or a regimen containing oxaliplatin, irinotecan, and 5-FU with or without leucovorin for treatment of advanced or metastatic disease, unless the patient refused such treatment. Up to two prior chemotherapeutic regimens are permitted.
3. Patients must have measurable disease including liver metastases >/= 2.0 cm amenable to percutaneous CT or U/S guided biopsy and must agree to undergo two liver biopsies.
4. Minimum of three weeks since any major surgery, radiation, or systemic anticancer therapy.
5. Any clinically significant residual adverse events from any prior anticancer therapy must have resolved to grade </= 1 or baseline as per the NCI Common Terminology Criteria for Adverse Events (CTCAE) v4.0.
6. Age >/=18 years. Because no dosing or adverse event data are currently available on the use of gene therapy in patients < 18 years of age, children are excluded from this study.
7. ECOG performance status 0 or 1.
8. Adequate hematologic, hepatic and renal parameters: leukocytes >/= 3,000/microliter, absolute neutrophil count >/= 1,500/microliter, platelets >/= 100,000/microliter, hemoglobin >/= 9g/dL, total bilirubin </= 1.5 mg/dL, AST and ALT </= 3 x upper limit of normal (ULN) for subjects with documented liver metastases; AST and ALT </= 2.5 x ULN for subjects without evidence of liver metastases, creatinine </= 1.5 mg/dL and calculated creatinine clearance of >/= 60 mL/min.
9. PT/PTT are within normal limits.
10. Women of childbearing potential must have a negative pregnancy test (serum or urine) within 14 days prior to treatment. Women must be surgically sterile or have been amenorrheic for at least 12 months to be considered of non-childbearing potential.
11. Women of childbearing potential and men must agree to use double barrier contraception prior to study entry and continuing for 30 days after the last dose of study drug.
12. Signed written informed consent/authorization form.

Exclusion Criteria:

1. Prior treatment with any investigational drug within the preceding 3 weeks of Cycle 1, Day 1.
2. Uncontrolled brain or leptomeningeal metastases, including patients who continue to require glucocorticoids for brain or leptomeningeal metastases (Brain imaging studies are not required if the patient does not have a history of brain metastases and has no neurological signs or symptoms).
3. Other malignancies within the past 3 years of Cycle 1, Day 1 except for adequately treated carcinoma of the cervix or basal or squamous cell carcinomas of the skin.
4. Patients who have any known severe and/or uncontrolled medical conditions or other conditions that could affect their participation in the study.
5. A known history of HIV seropositivity.
6. Women who are pregnant or breast feeding.
7. History of MI within 6 months of Cycle 1, Day 1, angina, history of arrhythmias on active therapy, patients with LV ejection fraction </= 50%.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-03; Primary Completion 2017-03 (Estimated); Study Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) of BikDD Nanoparticle in Patients with Advanced Pancreatic Cancer | Weekly during 28 day cycles
  The maximum tolerated dose (MTD) is defined as the maximal achievable dose level at which < 1/6 enrolled patients experiences dose-limiting toxicity.
Dose-Limiting Toxicity (DLT) | Continuously during 28 day cycles
  Dose-limiting toxicity (DLT) defined as:
  Any ≥ grade 3 hematologic and non-hematologic toxicity as per NCI CTCAE v. 4.0 with the following exceptions:
  1. Grade 3 or 4 lymphopenia unless persistent for >14 days or associated with single oral temperature of >38.3°C (101°F) or temp > 38°C (100.4°F) measured on two separate occasions one hour apart.
  2. Adverse events (Grade 3 or greater) for which a clinical cause unrelated to study drug is evident will not be considered DLTs. These will include: obstructive jaundice from stent occlusion, narcotic-induced constipation if symptom is present prior to study enrollment, anorexia or cachexia if present prior to study enrollment.
  3. Delay of Dose > 14 days due to toxicity.

CONTACTS AND LOCATIONS:
Overall Officials: Milind Javle, MD, Study Chair — M.D. Anderson Cancer Center

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org